CLINICAL TRIAL: NCT05771844
Title: Home Sleep Therapy System for Mild Cognitive Impairment
Brief Title: Home Sleep Therapy for Older Adults With MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brain Electrophysiology Laboratory Company (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R44AG077965 (NIH); 1R44AG077965-01A1 (NIH)
Record Dates: First submitted 2023-02-24; First posted 2023-03-16 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment; Sleep; Transcranial Electrical Stimulation; Machine Learning; Memory
Keywords: Slow Wave Sleep; NREM N3 Sleep
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: During Phase I of the study, all participants receive the same amount of TES stimulations, but in randomized order (stimulation either on the second night or the last night of Phase I). All participants receive stimulation and placebo in Phase II on a daily basis for up to two weeks at a time. The order participants receive placebo or treatment in the two week blocks are randomized.
Masking Description: All participants receive same amount of TES stimulations over the course of the study, but they are blind to which night or blocks of 2 weeks they receive the stimulation in Phases I and II of the study (stimulation either on the second night or the last night of Phase I and stimulation on either the first or last block of 2 weeks in Phase II).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Deep Sleep Enhancement with TES (Experimental): Transcranial Electrical Stimulation, 0.5 Hz sine wave, 0.5 mA, between frontal (frontopolar and inferior lateral frontal) and posterior (mastoid and occipital) electrodes.
  Interventions: Device: Transcranial Electrical Stimulation

INTERVENTIONS:
Device: Transcranial Electrical Stimulation — Oscillating electrical current
  Other Names: SleepWISP (Wireless Interface Sensor Pod)

SUMMARY:
The goal of this clinical trial is to learn about the ability of non-invasive brain stimulation during sleep to enhance people's deep sleep and its potential benefit on memory in people with mild cognitive impairment via home use sleep therapy device (SleepWISP) as well as learn about biomarkers associated with Alzheimer disease (AD). The clinical trial aims to answer the following main questions:

1. Whether the non-invasive transcranial electrical stimulation (TES) delivered by SleepWISP could provide short-term enhancement of deep sleep in a single night in the target population.
2. Whether TES delivered by SleepWISP could enhance deep sleep over multiple nights in the target population.
3. Whether enhance on deep sleep could improve memory performance in the target population.

Participants will be asked to wear non-invasive and painless devices that record their brain activity during sleep along with an actigraphy watch that measures their movement throughout the day. In addition, blood samples or nasal swab assays will be collected from participants multiple times during the study.

DETAILED DESCRIPTION:
The purpose of the present research is to evaluate the ability of non-invasive transcranial electrical stimulation (TES) during slow-wave sleep (SWS) to enhance this stage of sleep for people with mild cognitive impairment (MCI). A previous study of the investigators have demonstrated, in a pilot study, that TES can acutely (i.e., immediately after TES) increase SWS duration in healthy people. In the present proposal, the investigators aim to replicate and extend the pilot findings in seniors with MCI. It is evidenced that decline in SWS duration with aging is associated for memory impairment in seniors, which also creates risk for Alzheimer disease (AD). At the same time as conducting TES to enhance SWS sleep in seniors with MCI, the investigators also aim to explore changes in biomarkers associated with AD, including Aβ40 and Aβ42.

The investigators propose to conduct a sleep study using the Brain Electrophysiology Laboratory (BEL) company's Sleep WISP device (described in detail below). The Sleep WISP device is made up of three components: 1) 16-channel EEG amplifier with transcranial electrical stimulation (TES) capabilities, 2) a 16-channel EEG headband and 3) a small portable computer.

All participants will be provided a Sleep WISP device. Participation in the study requires that participants use the Sleep WISP when they sleep. As participants sleep, their sleep EEG will be measured and automatically scored by the computer to determine stage of sleep. When SWS is detected, low-level current (.5-1 mA total) will be applied through pre-set electrodes (four on the forehead and four at base of back of head). These electrodes were used in our pilot study, showing that current applied through these electrodes during SWS is able to increase total SWS sleep duration.

To evaluate the efficacy of the system, BEL will use a small, exploratory pilot sample of 10 employees and staff members to run the testing in Eugene, Oregon. After the 10 pilot subjects at BEL with employees and staff and prior to the main study, the protocol and system will be tested with older adults at each of the Wake Forest area (Winston-Salem, North Carolina) and Portland-Eugene surrounding area (Oregon) as pilot sub-studies for device usability feedback with seniors. These pilot subjects will only take part in the acute portion of the parent sleep study, where the first night is acclimation (no TES), the second night is TES or sham, and then a week later, they get TES or sham, for a total of three nights for the pilot studies. This pilot study does not include the PAVL memory test.

The greater study is divided into two phases.

Phase I involves up to nine sleep sessions. The first session is a baseline/acclimation session. In the first session, participants will use the Sleep WISP device to passively record sleep EEG (no TES) as baseline. The second session is performed the night following the baseline session with randomized experiment condition (either placebo or active TES session). Participants will be blinded for what condition they receive. The final session will occur one week after the second session to receive the opposite experiment condition to the second session. In the week between the second and final sessions, participants will be asked to wear the device at night to record their EEG. During this period, there will be no TES stimulation.

Phase II of the study can begin as early as the night following the completion of Phase I. To participate in Phase II participants do not need to have participated in Phase I. Phase II will follow a repeated-measures placebo-controlled design across six weeks. An equal number of participants without MCI (control group) and with MCI (experimental group) will be enrolled. Following screening and thorough training, participants will wear the WISP device for 2 weeks and receive either sham or treatment TES every night. A 2 week washout period where participants do not use the device will follow. Finally, participants will receive the remaining condition (sham or treatment) each night of the last 2 weeks of participation. Participants will also be asked to wear an actigraphy watch that measures sleep parameters based on movement each night in Phase II. A trained phlebotomist will collect blood samples or nasal swab assays from participants before and after each condition (sham and treatment; 4 total measurements) for Aβ detection.

In both Phases I and II, prior to sleep, participants will be presented with a paired-associate verbal learning (PAVL) task. Participants will be required to learn the list of words, to a pre-specified performance criterion. After waking from sleep in the morning, participants will be tested with the same list, to assess retention of the previously learned materials.

In our previous TES study of SWS enhancement, the investigators were able to show that SWS can be enhanced immediately (short-term/acute) after TES. The study was performed in the BEL sleep lab. Phase I of the proposed new study will extend the previous pilot study results by using Sleep WISP device as participants with MCI sleep at home, which will allow us to support home monitoring and acute treatment of disordered sleep for adults with MCI. Phase II will assess whether SWS modulation over multiple nights will produce cumulative enhancement of SWS in adults with MCI. In both study phases, the investigators will also evaluate the cognitive consequences, specifically declarative memory, of enhancing SWS.

Aim 1: Phase I aims to replicate our previous study (acute/short-term enhancement of SWS and safety/feasibility) in seniors with MCI with the sleep WISP device.

Aim 2: Phase II aims to assess the ability of TES to cumulatively enhance SWS over multiple sessions in seniors with MCI compared to healthy controls.

Aim 3: Evaluate SWS quality on a declarative memory task in older adults with MCI.

ELIGIBILITY:
Inclusion Criteria:

* For participant with Amnestic MCI, the inclusion age range is 55-85 years old.
* For healthy volunteers without MCI, the inclusion age range is 40-80 years old.

Exclusion Criteria:

* History of seizures
* History of epilepsy
* History of mod/severe brain injury or trauma (including neurosurgery)
* History or presence of significant neurological disease such as Parkinson
* History of Electroconvulsive Therapy (ECT)
* Presence of severe insomnia
* Presence of untreated sleep apnea
* Presence of severe anxiety or depression
* Medications that may affect the EEG
* History of stroke
* Sensitivity or allergy to lidocaine or silver
* Presence of active suicidal ideation
* Presence of metal in head or implants or medication infusion device
* Pregnancy
* Adverse reaction to TMS

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Device Usability | Collected each day they use the Sleep WISP system, for three sessions over 10 days during Phase I of the study.
  Criteria for success: the prototype is safe for all participants, and it is usable at home by 80% of adults with MCI. Specific outcome ratings (5-point Lickert scale) will be obtained for (1) ability to clean the device, (2) ability to apply the device, (3) ability to turn on the tablet (launching the dedicated software); (4) ability to start treatment; (5) ability to complete treatment.
Duration of N3 Sleep | Measured during the nights of sleep (typically 8 hours) across both phases of the study
  Duration in minutes of N3 sleep
Percentage of N3 Sleep | Measured during the nights of sleep (typically 8 hours) across both phases of the study
  Percentage of the night's sleep spent in N3

SECONDARY OUTCOMES:
Memory Performance; Paired-Associates Verbal Learning (PAVL) | Measured at the beginning as baseline, then once weekly over the course of study, and then once on the last day of the study, for a total of up to 7 times.
  10 pairs of unrelated, neutral-valence nouns are learned each night before sleep. Participants are tested in the morning when an online program provides the first word of the pair and they type in the second word that went with it (cued recall). More accurately recalled pairs of words (0-10 pairs) indicates better memory performance.
Beck Depression Inventory (BDI) | Measured at the beginning as baseline, then once weekly over the course of study, and then once on the last day of the study, for a total of up to 7 times.
  Assessment of psychiatric symptomatology; 21-item self-reported inventory that measures symptoms of depression. Responses are weighted and a higher score (1-40) indicates higher levels of depression.
Beta Amyloid Excretion Blood Sample or Nasal Swab Assay | Collected on the first day of Phase II of the study, and then the end of each week in Phase II, for a total of up to 7 times.
  Collected for exploratory analysis on biomarkers associated with Alzheimer's disease and treated with an anticoagulant, plasma isolated and stored at -80 until Aβ detection. Aβ40 and 42 detection will be performed using a commercially-available immunoassay (Innotest, Fugirebio).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Wake Forest University, Winston-Salem, North Carolina
  - Brain Electrophysiology Laboratory Company, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: Undecided